CLINICAL TRIAL: NCT05168072
Title: Weight Loss Effects of Mobile Health Application in Obesity Multidisciplinary Outpatient
Brief Title: Weight Loss Effects of M-health App in Obesity Multidisciplinary Outpatient Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: obesity2021
Record Dates: First submitted 2021-12-01; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Obesity; m-Health; NAFLD
Keywords: obesity; NAFLD; m-Health
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-Health (Experimental): participants receive conventional outpatient obesity management assisted with m-Health APP
  Interventions: Device: m-Health app; Other: conventional outpatient obesity management
- conventional (Active Comparator): participants receive conventional outpatient obesity management
  Interventions: Other: conventional outpatient obesity management

INTERVENTIONS:
Device: m-Health app — M-Health app is used to set weight loss targets and record body weights online. Participants learn the calories they consumed by using the m-Health APP and follow the APP for physical exercise
  Arms: m-Health
Other: conventional outpatient obesity management — Diet and exercise guidance

SUMMARY:
This is a randomized, open, controlled, single-center trial to identify the weight loss effects of adding mobile health application in obesity multidisciplinary outpatient clinic.

DETAILED DESCRIPTION:
This is a randomized, open, controlled, single-center trial to identify the weight loss effects of adding mobile health application in obesity multidisciplinary outpatient clinic.

The team of obesity multidisciplinary outpatient clinic includes endocrinologists, dietitians, and exercisers. The endocrinologist assesses the patients' conditions, manages the patients, and decides on appropriate medications. Dietitians participate in dietary propaganda and education, and develop personalized diet prescriptions. Exercisers conduct behavior and exercise propaganda, and issue personalized exercise prescriptions. Patients in the experimental group combine m-Health APP with routine obesity clinic management. The m-Health APP could help patients set weight loss targets, record body weights online, learn the calories they consumed in real time, and exercise based on the prescriptions suggested by the exercisers.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years old;
* 24kg/m^2 ≤ BMI < 37.5kg/m^2;
* Proficient in using mobile applications;
* Agree to sign the informed consent

Exclusion Criteria:

* secondary obesity (such as hypothyroidism, Cushing's syndrome, hypothalamic obesity or long-term use of obesity-causing drugs, etc.);
* Patients with chronic diseases that require special diet and affect exercise;
* Patients suffering from severe liver, kidney or heart dysfunction;
* Patients with a history of malignant tumor;
* Pregnant or lactating women;
* Low level of education or illiteracy;
* Inability, unwillingness, or refusal to comply with study requirements (including lifestyle adjustments, follow-up, and subject duties)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in weight loss | 12 weeks
  changes in body weight from baseline were observed after 12 weeks of treatment intervention
Changes in Nonalcoholic fatty liver disease | 12 weeks
  Changes in Nonalcoholic fatty liver disease (hepatic fibrosis index and liver fat attenuation parameters measured by Fibro touch) after 12 weeks of treatment

SECONDARY OUTCOMES:
Changes in body mass index (BMI(kg/m^2)=body weight(kg)/height(m^2)) of subjects | 12 weeks
  All 40 subjects of each group would be evaluated by changes in body mass index ( BMI(kg/m^2)=body weight(kg)/height(m^2)) after 12 weeks treatment
Changes in serum triglycerides, total cholesterol, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol | 12 weeks
  The changes in serum triglycerides, total cholesterol, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol would be measured at the beginning and the end.
Changes in serum alanine aminotransferase, aspartate aminotransferase and glutyltranspeptidase | 12 weeks
  The changes in serum alanine aminotransferase, aspartate aminotransferase and glutyltranspeptidase would be measured at the beginning and the end.

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD,PhD, Principal Investigator — the Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China